CLINICAL TRIAL: NCT01695551
Title: Assessment of Intracardiac and Surgace Electrogram Characteristics Correlated to Brain Perfusion and Hemodynamic Stability in Patients Undergoing Radiofrequency Ablation of Ventricular Tachycardia
Brief Title: Brain Perfusion and Hemodynamic Stability in Patients Undergoing Radiofrequency Ablation of Ventricular Tachycardia
Status: Completed | Type: Observational
Sponsor: Dhanunjaya Lakkireddy, MD, FACC (Other)
Responsible Party: Sponsor-Investigator, Dhanunjaya Lakkireddy, MD, FACC, Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Other Study IDs: 13054
Record Dates: First submitted 2012-07-05; First posted 2012-09-28 (Estimated); Last update posted 2017-01-09 (Estimated); Status verified 2017-01

CONDITIONS: Ventricular Tachycardia
Keywords: Radiofrequency ablation; fast heart rhythm; ventricle; catheter ablation; ablation
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ventricular Tachycardia: Participants in cohort will have implantable defibrillators in-situ and are undergoing ablation procedure for ventricular tachycardia.
  Interventions: Other: Data Collection Forms

INTERVENTIONS:
Other: Data Collection Forms — Participants will be asked questions relating to pre-procedure items and be asked to complete an MMSE. Subjects receive standard of care surgery. Data collected from procedures before, during and after surgery.

SUMMARY:
Ventricular tachycardia (VT) is a life-threatening, fast heart rhythm that starts in the lower chambers of the heart (the ventricles). This fast heartbeat is caused by abnormal electrical pathways located in the heart tissue. A standard procedure called a catheter ablation has been used for several years to help correct these abnormal pathways and, in some cases, improve or even eliminate the ventricular tachycardia.

During a VT ablation it is routine to monitor your vital signs (blood pressure, heart rate, and oxygen saturation in your blood). If you choose to participate in this study we will also monitor your cerebral oximetry, the amount of blood flow and oxygen saturation to your brain during the ablation.

By doing this study, we hope to have a better understanding of patients' blood and oxygen flow to their brain during an episode of Ventricular Tachycardia (VT).

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Have implantable defibrillator in-situ and are undergoing ablation procedure for ventricular tachycardia

Exclusion Criteria:

* Patients who have been hypotensive with systolic blood pressure of < 80mm Hg prior to procedure
* Cerebral event as defined by Cerebrovascular Accident or Transient Ischemia Attack within six months prior to procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from those that visit University of Kansas Medical Center Cardiology clinics.
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2012-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Identify clinical, EKG and EGM characteristics of hemodynamically unstable VT | Change from Baseline to 24-48 hours after surgery
  The investigator will be evaluating the relationship of the oxygenation level of the brain during a Ventricular Tachycardia ablation.

SECONDARY OUTCOMES:
MMSE to determine cerebral function before and after VT ablation | 24 hours after surgery
  The use of the Mini-Mental Status Exam prior to the ablation will serve as a reference point and will be repeated 24 hours post exam.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, FACC, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical center, Kansas City, Kansas, United States